CLINICAL TRIAL: NCT04930848
Title: Efficacy of Aqueous Extract of Euphorbia Hirta (Dudhiya) in Improving Sleep Quality: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effectiveness of Aqueous Extract(Tea) of Euphorbia Hirta (Dudhiya) in Improving Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Zannatun Nahar Nuri (Other)
Responsible Party: Sponsor-Investigator, Dr. Zannatun Nahar Nuri, Principal Investigator, Hamdard University
Organization: Hamdard University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HUBREC/2021/09/01
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Poor Sleep Quality
Keywords: Sleep; Quality; Herbal; Euphorbia hirta; Dudhiya; Randomized

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Euphorbia hirta
  Interventions: Other: Euphorbia hirta (Dudhiya)
- Placebo Arm (Placebo Comparator): Terminalia arjuna and Terminalia bellerica
  Interventions: Other: PBO(Combined powder of Terminalia arjuna and Terminalia bellerica)

INTERVENTIONS:
Other: Euphorbia hirta (Dudhiya) — Duration of the intervention was 2 consecutive weeks or 14 days. In each evening, one teaspoon full (3gm) powder should be mixed with two cups of water and boiled. When it becomes half(one cup), have to add one teaspoon of sugar and drink it as tea.
  Arms: Intervention Arm
Other: PBO(Combined powder of Terminalia arjuna and Terminalia bellerica) — Duration of the intervention was 2 consecutive weeks or 14 days. In each evening, one teaspoon full (3gm) powder should be mixed with two cups of water and boiled. When it becomes half(one cup), have to add one teaspoon of sugar and drink it as tea.
  Arms: Placebo Arm

SUMMARY:
Sound sleep is needed for our overall health and optimum our productivity. Sleep quality affects people's work performance, mood, safety, and quality of life. Changing times and advancements in technology couples with altered lifestyles have taken a toll on human health. Poor sleep quality reduces short-term memory, cognitive abilities, and motor skills for all age groups. The high prevalence of poor sleep quality in every age group has triggered a growing worldwide demand for a safe, effective and easily available herbal cure. Studies shown that, E. hirta has sedative action. For this, I hypothesized that oral intake of aqueous extract (tea) of E.hirta is efficacious in improving sleep quality.

In this study I assessed the efficacy of aqueous extract (tea) of Euphorbia hirta (Dudhiya) in improving sleep quality in persons aged 20 to 50 years with self-reported sleep disturbance.

The main objective of the study is to assess the efficacy of oral intake of aqueous extract of E.hirta in improving sleep quality in terms of having regular sound sleep and freshness in the daytime work.

A total of 32 adults with poor sleep quality was recruited for this study and included both of male and female.

Duration of the study was 05 months and active participation of each participant was 2 consecutive weeks or 14 days.

Study area was included Dhaka, Narayanganj and Munshiganj districts and study center was Dr. Hakeem Md. Yousuf Harun Bhuiyan Hospital, Hamdard University Bangladesh.

DETAILED DESCRIPTION:
Background:

Sound sleep is needed for our overall health and optimum our productivity. Sleep quality affects people's work performance, mood, safety, and quality of life. Changing times and advancements in technology couples with altered lifestyles have taken a toll on human health. Poor sleep quality reduces short-term memory, cognitive abilities, and motor skills for all age groups. The high prevalence of poor sleep quality in every age group has triggered a growing worldwide demand for a safe, effective and easily available herbal cure.

Therefore, in this study I assessed the efficacy of aqueous extract (tea) of Euphorbia hirta (Dudhiya) in improving sleep quality in persons aged 20 to 50 years with self-reported sleep disturbance.

Objective of the Study:

The main objective of the study is to assess the efficacy of oral intake of aqueous extract(Tea) of E.hirta compared with placebo (PBO) in improving sleep quality in terms of having regular sound sleep and freshness in the daytime work.

Sample Size:

Literature review have shown that sample size were included 24, 25, , 60, 112, 165 and 258 participants in sleep disorder related study. However, prior study on Withania somnifera in insomnia and anxiety has shown that the mean of the Pittsburgh Sleep Quality Index at the baseline was 13.08 and Standard Deviation (SD) 1.51, post-treatment & after follow up it was 9.15 and SD 1.8372. Based on this mean and SD, the estimated enrollment of 5 per treatment group among those with poor sleep would provide the study with a statistical power of 95% (α = 0.05) and confidence interval of 95% to detect significant improvements in sleep quality. By using OpenEpi online calculator, my required sample size is 10. Due to chance of loss to follow up and placebo effect (5%), my inflated sample size is total number of 32 participants which is three times larger than estimated sample size.

Duration of Study:

Duration of study for each participant was 05 months days with "day one advertisement" for screening followed by randomization for the treatment. The duration of the active participation of each participant 2 consecutive weeks or 14 days.

Study area was included Dhaka, Narayanganj and Munshiganj districts and study centre was Dr. Hakeem Md. Yousuf Harun Bhuiyan Hospital, Hamdard University Bangladesh.

Methods:

Participants was recruited by using online and printed advertisement of the study. Advertisements was posted on the online page of dept. of public health as well as other faculties of Hamdard University Bangladesh. Printed advertisement was posted on notice board of different faculties of Hamdard University Bangladesh along with providing in-person. Advertisements was also posted on online social networking platforms (such as Facebook, Facebook groups, LinkedIn). The relevant study requirements with an email address and phone number was included in the advertisement.

Interested respondent was contact to the investigator, and he/she was invited to come to Dr. Hakeem Md. Yousuf Harun Bhuiyan Hospital, Hamdard University Bangladesh for assessing sleep quality by self-reported Pittsburgh Sleep Quality Index questionnaire and checking physical parameters (i.e. general appearance, height, weight, body mass index (BMI), pulse rate, body temperature, blood pressure and respiratory rate) as well. Participants who met eligible criteria along with Pittsburgh Sleep Quality Index (PSQI) global score equal or greater than 6, and above mentioned physical parameters were normal -enrolled in this study.

After enrollment, they were randomized (by third party) into two groups to receive either the intervention or the placebo for 2 consecutive weeks or 14 days. A Sleep Diary also provided to each participants and instructed to complete it every morning within one hour after wake up. Participants were got reminder for taking intervention tea and completing sleep diary regularly every 2/3 days interval.

After completing intervention period, Participants were fulfilled another Pittsburgh Sleep Quality Index questionnaire for post-intervention assessment, and also fulfilled Sleep Diary was collected.

The Pittsburgh Sleep Quality Index contains seven component scores are, where the total score ranges from 0 to 21 points (0-3 points for each component). Lower scores indicate better sleep status. The global score is also calculated, with scores > 5 used to classify participants as "poor sleepers" and scores ≤5 used to classify participants as "good sleepers".

The outcome measure will be assessed by the differences between pre and post-intervention Pittsburgh Sleep Quality Index global score as well as the percentage reduction in Pittsburgh Sleep Quality Index compared with placebo.

To evaluate Subjective Sleep Efficiency (sSE) during the period of oral intake of aqueous extract of the intervention or placebo from sleep diary.

An intention-to-treat analysis will be conducted for patients who have received intervention at least once. Data will be presented as mean±SD and percentage of reduction in the change of improving sleep quality with a 95% confidence interval and p=0.05. sSE also be evaluated as percentage. Difference between two means will be compared with independent two sample t-test.

Efficacy Assessment:

1. Difference of baseline and post intervention mean by PSQI compared with PBO
2. Comparison of sSE between 1st and 14th day of intervention period from sleep diary
3. Assess the % of reduction of PSQI global score

Data and Safety Monitoring:

To maintain the quality of this trial, data & safety monitoring will be conducted by Data & Safety Monitoring Board (DSMB). The members of the DSMB was included that individual who was not involved directly in this research. For this clinical trial, DSMB members was joined from the Faculty of Unani and Ayurvedic Medicine of Hamdard University Bangladesh.

Safety Assessment:

Safety assessment was obtained from the incidence and type of adverse events during study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 20 to 50 years old
2. Having poor sleep quality (the PSQI global score ≥6) according to preliminary sleep assessment
3. Self-reported no problems with communication, both visual and auditory (reading, writing, hearing and speaking)
4. Signed the voluntary informed consent form for the clinical trial
5. Live in Dhaka, Narayanganj or Munshiganj district.

Exclusion Criteria:

1. Has taken western and/or oriental medicine and/or therapy and/or dietary supplements in the past 2 weeks for sleep disorders such as insomnia before the preliminary screening
2. Has a severe neural or psychiatric disorder or a history of major neuropsychiatric disorder e.g. autism, learning disorder, and mental retardation
3. Has a hemorrhagic disease or anticoagulant intake
4. Has a serious physical disorder i.e. heart disease, diabetes, cancer etc
5. Has participated in any other clinical trial within a month of the screening date
6. Pregnancy and lactation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Change in the Pittsburgh Sleep Quality Index global score. It's total score ranges from 0 to 21. The global score > 5 used to classify participants as "poor sleepers" and scores ≤5 used to classify participants as "good sleepers". | 14 days
  Difference of baseline and post intervention mean by the Pittsburgh Sleep Quality Index compared with placebo. Difference between two means will be compared with independent two sample t-test.
  Assess the % of reduction of Pittsburgh Sleep Quality Index global score, Baseline to 14 days.
Change in Subjective sleep efficiency(sSE) | 14 days
  Comparison of Subjective sleep efficiency(sSE) between 1st and 14th day of intervention period from sleep diary.

CONTACTS AND LOCATIONS:
Overall Officials: Zannatun N Nuri, BAMS, Principal Investigator — MPH student, Hamdard University Bangladesh
Locations (1):
- Hamdard University Bangladesh, Munshiganj, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting 6 months after publication.
Access Criteria: Request by email.